CLINICAL TRIAL: NCT06135012
Title: Influence of Pancreatic Transection With Cavitron Ultrasonic Surgical Aspirator (CUSA) on Postoperative Pancreatic Fistula Incidence - a Prospective Randomised Controlled Trial: the PANCUT Study
Brief Title: Influence of Pancreatic Transection With CUSA on Postoperative Pancreatic Fistula Incidence (PANCUT)
Acronym: PANCUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230052
Record Dates: First submitted 2023-07-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic surgery; Pancreas transection; Postoperative complications; POPF
MeSH Terms: conditions — Pancreatic Fistula; Postoperative Complications | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transection with CUSA (Experimental): Transection of pancreatic tissue using cavitron ultrasonic surgical aspirator (CUSA) and using metal clips for closing small intraparenchymal blood vessels and pancreatic branch ducts.
  Interventions: Device: Cavitron ultrasonic surgical aspirator (CUSA)
- Transection with scalpel/stapler (Sham Comparator): Standard transection of pancreatic tissue with a surgical scalpel without selective closure of small blood vessels and branch pancreatic ducts (in pancreaticoduodenectomy).
  Interventions: Other: Scalpel

INTERVENTIONS:
Device: Cavitron ultrasonic surgical aspirator (CUSA) — Transection of pancreatic tissue with cavitron ultrasonic surgical aspirator (CUSA).
  Arms: Transection with CUSA
Other: Scalpel — Transection of pancreatic tissue with scalpel.
  Arms: Transection with scalpel/stapler

SUMMARY:
Objective: To compare the outcomes after elective pancreatic resections using cavitron ultrasonic surgical aspirator (CUSA) and selective closure of small blood vessels and branch pancreatic ducts versus surgical scalpel or stapler for the transection of pancreatic tissue.

Study design: A randomized controlled, single centre trial.

Study population: Two groups of 80 patients (160 in total) scheduled for elective open pancreaticoduodenectomy (PD) for any indication.

Intervention: Transection of pancreatic tissue with CUSA.

Control: Standard transection of pancreatic tissue with surgical scalpel (in PD) or stapler (in DP)

DETAILED DESCRIPTION:
Rationale: Postoperative pancreatic fistula (POPF) is one of the major causes of morbidity and mortality after pancreatic resections. There is no predominant surgical technique of pancreatic stump closure in distal pancreatectomy (DP) or formation of pancreaticojejunostomy in pancreaticoduodenectomy (PD) proven to prevent/lower POPF incidence. Cavitron ultrasonic surgical aspirator (CUSA) selectively removes tissue parenchyma, evading blood vessels and pancreatic ducts which could consequently be selectively ligated. Such technique could anull pancreatic juice drainage from branch ducts and provide better (skeletonised) view of the main duct to from an anastomosis (or to ligate it in DP) and thus lower the incidence of POPF formation.

Objective: To compare transection of pancreatic tissue with CUSA and selective closure of small blood vessels and branch pancreatic ducts with transection with surgical scalpel or stapler in elective pancreatic resections regarding the incidence of POPF.

Study design: A randomized controlled, single centre trial. The study protocol was designed according to the SPIRIT guidelines.

Study population: Two groups of 80 patients (160 in total) scheduled for elective open pancreaticoduodenectomy (PD) for any indication.

Intervention: Transection of pancreatic tissue with CUSA.

Control: Standard transection of pancreatic tissue with surgical scalpel (in PD).

Main study parameters/endpoints: Primary outcome is the incidence of POPF. Main secondary outcomes are intraoperative outcomes (such as blood loss and operative time), postoperative outcomes (such as complications, time to functional recovery and hospital stay).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more
* Patients capable of understanding the provided information about the study
* Patients with signed informed consent
* Planned elective pancreaticoduodenectomy for any indication

Exclusion Criteria:

* Patients aged less than 18
* Patient incapable of understanding the provided information about the study
* Pregnancy
* Previous surgical procedures on pancreas
* Immunosuppressive therapy
* Preoperative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula incidence | 30 days
  Evaluation and incidence of postoperative pancreatic fistula

SECONDARY OUTCOMES:
Postoperative septic complications | 90 days
  Intraabdominal collections, antibiotic treatment
Number of postoperative interventions | 90 days
  Percutaneous drain placement or reoperations
Hospital stay | 90 days
  Days in hospital
Volume of intraoperative blood loss | 1 day
  Blood loss during surgery
Operative time | 1 day
  Time spent for pancreas transection

CONTACTS AND LOCATIONS:
Overall Officials: David Badovinac, Principal Investigator — Department of Abdominal Surgery, University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hadzialjevic B, Zavrtanik Carni H, Petric M, Dokic M, Trotovsek B, Tomazic A, Badovinac D. Influence of pancreas transection with cavitron ultrasonic surgical aspirator (CUSA) on incidence of postoperative pancreatic fistula after pancreatoduodenectomy (PANCUT): study protocol for a randomised controlled trial. Trials. 2025 Jun 4;26(1):190. doi: 10.1186/s13063-025-08898-4. PMID 40462161